CLINICAL TRIAL: NCT07121634
Title: Cervical Ripening With Misoprostol Versus Isosorbide Mononitrate in Late-term Pregnancies: A Prospective Parallel -Arm Randomized Controlled Trial
Brief Title: Cervical Ripening With Misoprostol vs Isosorbide Mononitrate ; A Parallel -Arm Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raid M. Al-Ani (Other)
Responsible Party: Sponsor-Investigator, Raid M. Al-Ani, Professor, University Of Anbar
Organization: University Of Anbar (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Anbar
Record Dates: First submitted 2025-07-17; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cervical Ripening
Keywords: Misoprostol; Isosorbide Mononitrate; Pregnancy, Prolonged
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Misoprostol; isosorbide-5-mononitrate; Nitric Oxide Donors

STUDY DESIGN:
Intervention Model Description: Arm 1 Arm Title: Misoprostol Group Arm Type: Experimental
  Arm Description:
  Participants in this group received 25 µg of Misoprostol (Vagiprost; ADWIA Co/Egypt) administered vaginally every 4 hours, up to a maximum of 3 doses, for cervical ripening before induction of labor.
  Assigned Intervention:
  Drug Name: Misoprostol • Other Names: Vagiprost, synthetic prostaglandin E1 Arm 2 Arm Title: Isosorbide Mononitrate Group Arm Type: Active Comparator
  Arm Description:
  Participants in this group received 40 mg of Isosorbide Mononitrate (Monomack; Mack Pharmaceutics, Jordan) administered vaginally every 4 hours, up to 3 doses, as a nitric oxide donor agent for cervical ripening.
  Assigned Intervention:
  Drug Name: Isosorbide Mononitrate
  • Other Names: IMN, Monomack, nitric oxide donor
Who Masked: Outcomes Assessor
Masking Description: blinded assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol group (Experimental): Misoprostol Group Arm Type: Experimental
  Arm Description:
  Participants in this group received 25 µg of Misoprostol (Vagiprost; ADWIA Co/Egypt) administered vaginally every 4 hours, up to a maximum of 3 doses, for cervical ripening before induction of labor.
  Assigned Intervention:
  Drug Name: Misoprostol
  • Other Names: Vagiprost, synthetic prostaglandin E1
  Interventions: Drug: Misoprostol 25 µg Vaginal
- Isosorbide Mononitrate Group (Experimental): The Isosorbide Mononitrate group (n=40) were nitric acid donor cases applied to the posterior fornix prior to induction of labor. Isosorbide mononitrate (IMN) (Monomack; Mack Pharmaceutics; Jordan) in a vaginal dose of 40 mg was used every 4 hours (up to 3 doses).
  Interventions: Drug: Isosorbide Mononitrate

INTERVENTIONS:
Drug: Misoprostol 25 µg Vaginal — The Misoprostol group (n=40) were Misoprostol cases, a synthetic PGE1 in the form of vaginal tablets of 25 µg (Vagiprost; ADWIA Co/Egypt) applied locally to the posterior fornix every 4 hours for cervical ripening before induction of labor is started (up to 3-doses).
  Other Names: Cytotec Vagiprost PGE1 analogue
  Arms: Misoprostol group
Drug: Isosorbide Mononitrate — The Isosorbide Mononitrate group (n=40) were nitric acid donor cases applied to the posterior fornix prior to induction of labor. Isosorbide mononitrate (IMN) (Monomack; Mack Pharmaceutics; Jordan) in a vaginal dose of 40 mg was used every 4 hours (up to 3 doses).
  Women who scored a BS of > 6 from the assigned time were labelled as (1), after the passage of 40 hours, while those women whose BS was less than 6 were labelled (0) for construction of the Kaplan Meier curve for both groups.
  Other Names: IMN, Monomack, Nitric oxide donor
  Arms: Isosorbide Mononitrate Group

SUMMARY:
This randomized controlled trial compared misoprostol and isosorbide mononitrate (IMN) for cervical ripening in prolonged pregnancies. Low-risk women at 41+6 weeks gestation with an unfavorable cervix were randomized to receive either misoprostol or IMN. The primary outcome was the achievement of cervical ripeness (Bishop Score ≥6) within 40 hours.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the effectiveness and safety of misoprostol versus isosorbide mononitrate (IMN) for cervical ripening in prolonged pregnancies (≥41+0 weeks gestation). Favorable cervical status, reflected by a Bishop Score ≥6, is critical for successful vaginal delivery. Participants are low-risk pregnant women at 41+6 weeks with an unfavorable cervix. They are randomized to receive either 25 mcg of vaginal misoprostol or 40 mg of vaginal IMN, administered every 4 hours for up to 3 doses. Cervical status is assessed at regular intervals to determine the achievement of cervical ripening within 40 hours.

The primary outcome is the proportion of participants achieving a Bishop Score ≥6. Secondary outcomes include maternal parameters (labor progression, cesarean section rate, postpartum hemorrhage) and neonatal outcomes (Apgar scores, fetal heart rate tracing, and Doppler indices). The study aims to determine which agent more effectively facilitates cervical ripening and supports favorable delivery outcomes in late-term pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk primigravidae
* Singleton viable pregnancy
* Cephalic fetal presentation
* Confirmed gestational age ≥ 41+0/7 weeks
* Normal fetal growth pattern
* No signs of labor at the time of enrollment

Exclusion Criteria:

* High-risk pregnancies
* Body mass index (BMI) > 30 kg/m²
* History of unexplained fetal death
* Oligohydramnios or fetal distress
* Abnormal placentation
* Rh-negative status
* Pre-existing medical conditions or contraindications to labor induction or study drugs
* Fetal abnormalities
* Malpresentation or malposition
* Inadequate pelvimetry
* Participants who developed fetal distress or failed to progress during induction and required emergency cesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Ripening Success | Time Frame: Up to 40 hours post-intervention
  Proportion of participants achieving Bishop Score ≥6 within 40 hours after receiving Misoprostol or Isosorbide Mononitrate.
  Unit of Measure: Percentage of participants (%)

OTHER OUTCOMES:
Cesarean Section | during delivery
  Rate of Cesarean Section Proportion of participants who underwent cesarean delivery. Unit of Measure: Percentage of participants (%)
Postpartum Hemorrhage Unit of Measure: Number of participants | Delivery to 2 hours postpartum
  Number of participants with blood loss ≥500 mL during or within 2 hours after delivery.
abnormal fetal heart tracing during labor | during delivery
  number of fetuses who develop abnormal heart tracing
Neonatal Apgar Score <7 at 1 Minute Unit of Measure: Number of neonates | Time Frame: 1 minute post-delivery
  Description: Number of neonates with Apgar score <7 at 1 minute after birth.
Neonatal Apgar Score <10 at 5 Minutes | 5 minutes post-delivery
  Number of neonates with Apgar score <10 at 5 minutes after birth.
  Unit of Measure: Number of neonates

CONTACTS AND LOCATIONS:
Overall Officials: Wassan Nori, PhD, Principal Investigator — Al-Mustansiriyah University
Locations (1):
- Yarmouk, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No